CLINICAL TRIAL: NCT06380088
Title: Improving Motor Task Performance: Music and Verbal Encouragement as Catalysts - Highlights From Electromyographic Analysis
Brief Title: Improving Motor Skills: The Role of Music and Encouragement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita degli Studi di Genova (Other)
Responsible Party: Principal Investigator, Luca Puce, Principal Investigator, Universita degli Studi di Genova
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: VEM-DINOGMI-24
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: muscle fatigue; Neuromuscular Strategy; performance; sEMG; Motor recruitment; Motivation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Task with music (Experimental): Endurance isometric exercise performed to selected music.
  Interventions: Other: Isometric Task
- Task with verbal encouragement (Experimental): Endurance isometric exercise performed with verbal encouragement.
  Interventions: Other: Isometric Task
- Task without motivational feedback (Experimental): Task without motivational feedback.
  Interventions: Other: Isometric Task

INTERVENTIONS:
Other: Isometric Task — The exercise required participants to keep their arm flexed at a 90° angle while holding a dumbbell loaded to 80% of their 1RM (One Rep Max) in a supine position on the dominant side of the body for as long as possible.

SUMMARY:
This study used a randomised crossover design to analyse the effect of three different experimental interventions - i.e. standard conditions, music and verbal encouragement - on performance in an isometric endurance task, comparing results between untrained and trained individuals. The interval between each intervention was set at seven days. The outcome measures are muscle activity and fatigue, assessed by surface electromyography, and task duration.

Isometric endurance task requires participants to keep their arm flexed at a 90° angle while holding a dumbbell with a supine grip loaded to 80% of 1RM on the dominant side of the body. During execution, the back and head should remain in contact with a vertical wall, with the feet shoulder width apart and firmly planted on the floor. The bar is held with the dominant arm while the other arm remains in a neutral position close to the body. It is imperative to avoid any form of rocking or movement that would make it easier to maintain the position. The test officially begins when the bar is handed to the subject, who is already in the correct position, and ends as soon as the angle of the arm varies by more than five degrees from the starting position.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, candidates had to be in good general health, with no medical conditions that could interfere with their ability to perform the test safely and effectively. In addition, to be considered trained, participants had to have performed 150 minutes per week of vigorous-intensity aerobic physical activity, in addition to muscle-strengthening activities, on at least two days per week. Those who did not meet this standard were considered untrained.

-

Exclusion Criteria:

Exclusion criteria included a history of surgery to the arm, shoulder, or nearby areas that could limit the ability to perform the test. The use of medications that affect muscle function or pain perception was also a reason for exclusion, so that the test results could not be influenced by external factors.

-

Ages: 27 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Duration of the task | 60 seconds
  task duration expressed in seconds
Biceps Brachii muscle fatigue | 60 seconds
  time-course evolution of the median frequency of the power density spectrum (MF [Hz]) of the sEMG signal measured for Biceps Brachii muscle
Triceps Brachii muscle fatigue | 60 seconds
  time-course evolution of the median frequency of the power density spectrum (MF [Hz]) of the sEMG signal measured for Triceps Brachii muscle
Biceps Brachii activity | 60 seconds
  time-course evolution of the amplitude (Root Mean Square [microvolt]) of the sEMG signal measured for Biceps Brachii muscle
Triceps Brachii activity | 60 seconds
  time-course evolution of the amplitude (Root Mean Square [microvolt]) of the sEMG signal measured for Triceps Brachii muscle

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi di Genova, Genova, Italy

IPD SHARING:
Plan to Share IPD: No